CLINICAL TRIAL: NCT02644460
Title: Abemaciclib in Children With Newly Diagnosed Diffuse Intrinsic Pontine Glioma, and in Children With Recurrent and Refractory Solid Tumors Including Malignant Brain Tumors
Brief Title: Abemaciclib in Children With DIPG or Recurrent/Refractory Solid Tumors
Acronym: AflacST1501
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Thomas Cash, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00083793
Record Dates: First submitted 2015-12-15; First posted 2015-12-31 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Brain Tumor, Recurrent; Solid Tumor, Recurrent; Neuroblastoma, Recurrent, Refractory; Ewing Sarcoma, Recurrent, Refractory; Rhabdomyosarcoma, Recurrent, Refractory; Osteosarcoma, Recurrent, Refractory; Rhabdoid Tumor, Recurrent, Refractory
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Brain Neoplasms; Recurrence; Neuroblastoma; Sarcoma, Ewing; Rhabdomyosarcoma; Osteosarcoma; Rhabdoid Tumor | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stratum A (Experimental): Appropriate dose RT will be administered in 30-33 fractions over approximately 6 weeks for Stratum A patients. Treatment with abemaciclib (LY2835219) will start on the same day as RT and continue twice daily during and after RT for a maximum treatment duration of 2 years. Investigators plan to treat a maximum of 4 cohorts of research participants (dosage levels 1, 2, 3, and 4) with escalating doses of abemaciclib (LY2835219) starting with dose level 1 (80% of adult dose). A cycle is defined as 28 days and the first 6 weeks of therapy will constitute the dose-limiting toxicity (DLT)-evaluation period. Participants must take abemaciclib by mouth as intact capsules.
  Interventions: Drug: Abemaciclib
- Stratum B - enrollment is closed for this study arm (Experimental): Abemaciclib (LY2835219) will be administered orally on a twice daily basis continuously for 28 days, which defines one cycle. The maximum treatment duration will be 2 years. Investigators plan to treat a maximum of 4 cohorts of research participants (dosage levels 1, 2, 3, and 4) with escalating doses of abemaciclib starting with dose level 1 (80% of adult dose). Dose escalation will be independent of Stratum A escalation. A cycle is defined as 28 days and the first 4 weeks of therapy will constitute the DLT-evaluation period. Participants must take abemaciclib by mouth as intact capsules.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib
  Other Names: LY2835219

SUMMARY:
This is a Phase I clinical trial evaluating abemaciclib (LY2835219), an inhibitor of cyclin dependent-kinases 4 and 6 (Cdk 4/6) in children and young adults with newly diagnosed diffuse intrinsic pontine glioma (DIPG) (Stratum A) and in relapsed/refractory/progressive malignant brain (Grade III/IV, including DIPG; MBT) and solid tumor (ST) patients (Stratum B).

DETAILED DESCRIPTION:
Stratum A- Appropriate dose RT will be administered in 30-33 fractions over approximately 6 weeks for Stratum A patients. Treatment with abemaciclib (LY2835219) will start on the same day as radiation therapy (RT) and continue twice daily during and after RT for a maximum treatment duration of 2 years. Investigators plan to treat a maximum of 4 cohorts of research participants (dosage levels 1, 2, 3, and 4) with escalating doses of abemaciclib (LY2835219) starting with dose level 1 (80% of adult dose). A cycle is defined as 28 days and the first 6 weeks of therapy will constitute the dose-limiting toxicity (DLT)-evaluation period. Participants must take abemaciclib by mouth as intact capsules.

Stratum B (no longer enrolling) - Abemaciclib (LY2835219) will be administered orally on a twice daily basis continuously for 28 days, which defines one cycle. The maximum treatment duration will be 2 years. Investigators plan to treat a maximum of 4 cohorts of research participants (dosage levels 1, 2, 3, and 4) with escalating doses of abemaciclib starting with dose level 1 (80% of adult dose). Dose escalation will be independent of Stratum A escalation. A cycle is defined as 28 days and the first 4 weeks of therapy will constitute the DLT-evaluation period. Participants must take abemaciclib by mouth as intact capsules.

Enrollment for Stratum B closed December 27, 2018.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Patient must have measurable or evaluable disease.
* Age must be ≥ 2 years and < 25 years
* Body surface area (BSA) ≥ 0.5 m^2
* Lansky (for participants ≤ 16 years) or Karnofsky (for participants > 16 years) performance score ≥ 40 at the time of study enrollment
* Adequate organ function at the time of study enrollment as follows:

  * Bone marrow: Absolute neutrophil count (ANC) ≥ 1,000/μL, platelet count ≥ 75,000/μL (transfusion independent for ≥ 7 days), hemoglobin concentration ≥ 8g/dL (may be transfused)
  * Patients with bone marrow metastatic disease who do not meet the above criteria will be eligible to enroll in the study with the following count criteria. These patients will not be evaluable for hematologic toxicity or hematologic DLT.

    * ANC > 750/μL within 7 days prior to first dose of abemaciclib
    * Platelet count > 50,000/μL (may receive platelet transfusions) within 7 days prior to first dose of abemaciclib
    * Hemoglobin ≥ 7.5 g/dL (may receive red blood cell (RBC) transfusions) within 7 days prior to first dose of abemaciclib
  * Renal: Normal serum creatinine concentration based on age or glomerular filtration rate (GFR) > 70 ml/min/1.73m^2
  * Hepatic: Total bilirubin concentration < 1.5x the institutional upper limit of normal for age; serum glutamic pyruvic transaminase (SGPT) < 10x the institutional upper limit of normal for patients on Stratum A. Stratum B patients must have SGPT < 4x the institutional upper limit of normal.
  * Cardiac: Adequate cardiac conductivity with corrected Q-T interval (QTC) of < 450 ms on screening ECG.
* Female research participants of childbearing age must not be pregnant as confirmed by a serum or urine pregnancy test within 1 week of start of treatment. Participants must not be breast-feeding.
* All patients should submit an archival tumor biopsy specimen (collected at diagnosis or relapse). Patients who have no tumor tissue available may be permitted to participate after discussion with the principal investigator.
* Males or females of reproductive potential may not participate unless they have agreed to use two effective contraceptive methods. Abstinence in a non-sexually active child will be sufficient birth control.

Inclusion Criteria for Stratum A (Newly Diagnosed DIPG)

* Diagnosis of DIPG or high-grade glioma originating from the brainstem
* Participants have had no previous treatment except corticosteroid use.

Inclusion Criteria for Stratum B (Recurrent/refractory/progressive MBT (including DIPG) or ST) - Stratum B is closed to further accrual of participants

* Patients must have radiologic evidence of recurrent, refractory or progressive malignant central nervous system (WHO Grade III or IV) or solid tumor. For patients with radiologic features of DIPG histologic confirmation of diagnosis is not required though biopsy is suggested if clinically indicated.
* Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration.
* Patients who are on dexamethasone must be on a stable or decreasing dose for at least one week prior to registration.
* Patients must have fully recovered from the acute toxic effects of chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
* Myelosuppressive chemotherapy: Patients must have received their last dose of known myelosuppressive anticancer chemotherapy at least 21 days prior to study registration or at least six weeks if nitrosourea. At least two weeks must have lapsed if patients received lower dose oral etoposide (50 mg/2) without experiencing evidence of myelosuppression (i.e. neutropenia or requiring transfusion with blood products)
* Biologic agent: Patient must have recovered from any toxicity potentially related to the agent and received their last dose of the biologic agent ≥ 7 days prior to study registration.
* Monoclonal antibody treatment: At least three half-lives must have elapsed prior to registration.
* Radiation: Patient has received radiation therapy prior to study registration. Patients must have had their last fraction of local irradiation to the primary tumor ≥ 3 months prior to registration, their last fraction of craniospinal irradiation (>24Gy) or total body irradiation > 3 months prior to registration or > 6 wks for therapeutic doses of metaiodobenzylguanidine (MIBG). Patient has not received focal irradiation for symptomatic metastatic sites within 14 days prior to registration.
* Bone Marrow Transplant: Patient must be ≥ 3 months since high dose chemotherapy and peripheral blood stem cell rescue prior to registration.
* Autologous stem cell transplant following myeloablative therapy within 3 months prior to the first dose of abemaciclib or prior allogeneic stem cell transplant at any time. Patients who received stem cell reinfusion following non-myeloablative therapy are eligible once they meet peripheral blood count criteria.
* Growth factors: Patients must be off all colony forming growth factors(s) for at least 1 week prior to registration (filgrastim, sargramostim, erythropoietin) and at least 2 weeks for long-acting formulations (e.g. Neulasta).

Exclusion Criteria:

* Patients with uncontrolled infection
* Patients with any concomitant significant medical illness that in the investigator's opinion cannot be adequately controlled with appropriate therapy, or that would impair the evaluation of side effects related to this treatment, alter drug metabolism or the tolerance to this treatment
* Patients receiving any other anticancer or investigational drug therapy
* Prior therapy with abemaciclib
* Known mutation of Rb in tumor tissue
* Prior history of QTC prolongation or QTC>450 ms on screening ECG.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Abemaciclib Maximum Tolerated Dose (MTD) for Diffuse Intrinsic Pontine Glioma (DIPG) | Week 6
  The maximum dose of abemaciclib tolerated in participants with newly diagnosed diffuse intrinsic pontine glioma (DIPG).
Abemaciclib Maximum Tolerated Dose (MTD) for Recurrent/Refractory Solid Tumors | Week 6
  The maximum dose of abemaciclib in participants with recurrent/refractory solid tumors, including malignant tumors of the brain and spine.
Pharmacokinetics (PK): Predose Concentration (Cmin) of Abemaciclib | Cycle 1 to End of Study (up to two years)
Pharmacokinetics (PK): Maximum Concentration (Cmax) of Abemaciclib | Cycle 1 to End of Study (up to two years)
Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of Abemaciclib | Cycle 1 to End of Study (up to two years)

SECONDARY OUTCOMES:
Number of participants with adverse events | End of study (Up to two years)
  The number of participants who experience adverse events.
Number of hematological toxicities | End of study (Up to two years)
  The number of hematological toxicities observed throughout the study among participants.
Number of non-hematological toxicities | End of study (Up to two years)
  The number of non-hematological toxicities observed throughout the study among participants.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cash, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Egleston, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Scottish Rite, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903